CLINICAL TRIAL: NCT07379801
Title: The Musculoskeletal System During Puberty in Dancers With Scoliosis, and the Effect of an Exercise Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Gali Dar, PHD, Prof., University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 034/26
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Development, Adolescent
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 2 groups - dancers with scoliosis will be randomly assigned to either a three-month targeted exercise program or a control group continuing regular training.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- excercise (Experimental): exercises for strengthening
  Interventions: Other: exercise
- control (No Intervention): regular activity

INTERVENTIONS:
Other: exercise — exercise for strengthening core muscles
  Arms: excercise

SUMMARY:
assessment of the musculoskeletal system will be performed twice a year, for three years of young dancers

DETAILED DESCRIPTION:
Objectives: To examine musculoskeletal system characteristics in female dancers with and without scoliosis throughout the pubertal period, and to evaluate the effect of a targeted preventive exercise program.

Methods: Up to 140 female dancers aged 11-16 will be recruited for a two-phase study:

Phase A: a two-year longitudinal study with four assessment time points. . At each time point, participants will complete a comprehensive assessment including: anthropometric measurements (height and weight), sexual maturation status (Tanner scale), scoliosis assessment (Adam's forward bend test, scoliometer measurements, Scoliosis Research Society-22 questionnaire), bone strength (quantitative ultrasound using a Speed of Sound [SOS] device), abdominal and back muscle morphology (ultrasound imaging), hip muscle strength (handheld dynamometry), hip range of motion (goniometry), dynamic balance (Y Balance Test), and flexibility (Beighton score). In addition, participants will complete a demographic questionnaire and an injury surveillance questionnaire.

Phase B : an intervention study in which dancers with scoliosis will be randomly assigned to either a three-month targeted exercise program or a control group continuing regular training. Outcomes will be assessed post-intervention and at one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female dancers aged 11-16 years who dance at least three times per week and whose parents have provided informed consent.
* Dancers who have participated in at least three weekly hours of classical ballet during the year preceding the study and during the study year.
* A minimum of two years of experience in classical ballet training.
* Dancers without underlying medical conditions, not taking medications, and with no history of orthopedic surgery.
* dancers diagnosed during the study with mild to moderate scoliosis who are not under medical follow-up requiring active orthopedic or surgical treatment.

Exclusion criteria:

- Dancers who are taking medications, are not in good health, have underlying medical conditions, or have undergone any orthopedic surgery.

Ages: 11 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — females dencers
Enrollment: 140 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
ultrasound for muscle thickness | baseline, twice a year for 2 years
  ultrasound assessment of back and abdominal muscles in rest and contraction - thickness in mm
muscle strength test | baseline, twice a year for 2 years
  hand held dynamometer assessment hip muscles
range of motion | baseline, twice a year for 2 years
  goniometer assessment for lower extremities joints
bone strength | baseline, twice a year for 2 years
  tibia bone strength assessment using Sunlight MiniOmni Ultrasound Bone Sonometer
maturation status | baseline, twice a year for 2 years
  Tanner scale 0-5 scale. higher score represent greater maturation status
scoliosis | baseline, twice a year for 2 years
  Adam's tests and scoliometer
flexibility | baseline, twice a year for 2 years
  Beighton score. 0-9 scale when higher score represent hyper flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, PhD, Principal Investigator — University of Haifa
Locations (1):
- Haifa University, Department of PHysical Therapy, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will be shared with other researchers upon reasonable request and in coordination with the principal investigator, subject to ethical approval and data use agreements.

REFERENCES:
- [Background] Dar G, Elbaz L, Vilnai T, Ben-Zvi D, Grinstein M, Steinberg N. Hyperlaxity and low bone mass predispose young female gymnasts to develop scoliosis suspected status. Sci Rep. 2025 Jul 2;15(1):22827. doi: 10.1038/s41598-025-05895-0. PMID 40594709